CLINICAL TRIAL: NCT01219881
Title: A Randomized, Double-Blind, Double-Arm Trial Comparing Desflurane to Sevoflurane for the Effect on Recovery Time in Patients Undergoing Urological Cystoscope Surgery Under General Anesthesia With a Laryngeal Mask Airway (LMA)
Brief Title: Comparing Desflurane to Sevoflurane for the Effect on Recovery Time in Patients Undergoing Urological Cystoscope Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2010H0174
Record Dates: First submitted 2010-09-27; First posted 2010-10-13 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Cystoscopes; Baxter Anaesthesia Brand of Desflurane; Sevoflurane
Keywords: desflurane; sevoflurane
MeSH Terms: interventions — Desflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desflurane (Active Comparator): Comparing the effect on recovery time in patients undergoing urological cytoscope surgery under general anesthesia with a laryngeal mask airway (LMA) using Desflurane.
  Interventions: Drug: Desflurane
- Sevoflurane (Active Comparator): Comparing the effect on recovery time in patients undergoing urological cytoscope surgery under general anesthesia with a laryngeal mask airway (LMA) using Sevoflurane.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Desflurane — 5.4 to 7.4% desflurane
  Arms: Desflurane
Drug: Sevoflurane — 1.4 to 2.5% Sevoflurane
  Arms: Sevoflurane

SUMMARY:
This is a single-center, prospective, randomized, double-blind, double-arm trial including 68 subjects scheduled to undergo urological cystoscope surgeries under general anesthesia (GA) with intubation through a laryngeal mask airway (LMA) at The Ohio State University Medical Center (OSUMC). Double blinding will be based on both the subject and the research staff being unaware of which trial arm the subject is randomized into. Eligible subjects that provide voluntary and written informed consent will be included in this study.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, double-blind, double-arm trial including 68 subjects scheduled to undergo urological cystoscope surgeries under general anesthesia (GA) with intubation through a laryngeal mask airway (LMA) at The Ohio State University Medical Center (OSUMC). Double blinding will be based on both the subject and the research staff being unaware of which trial arm the subject is randomized into. Eligible subjects that provide voluntary and written informed consent will be included in this study.

Day -14 to 0

Subjects will undergo screening procedures up to 14 days prior to administration of study treatment. The research staff will collect the subjects' medical history (including reason for surgery, scheduled surgical procedure, anesthesia modality, and scheduled surgery length), demographics (including gender, age, and race), allergies, history of smoking, history of alcohol or drug abuse, medications, history of postoperative nausea and vomiting (PONV), and history of motion sickness. A physical examination will also be performed at this time.

Day 0

Upon enrolment, subjects will be randomly assigned in a 1:1 ratio, from a pre-determined randomization schedule, by the research pharmacist to one of two anesthetic treatment groups: Anesthesia maintained under desflurane or anesthesia maintained under sevoflurane.

Prior to surgery, a urine or serum pregnancy test will be performed and vitals will be collected. Subjects' baseline pain and nausea will be assessed using an eleven point numeric rating scale (NRS-11)15, where 0 is equivalent to none and 10 is equivalent to severe, prior to entering the operating room (OR).

Cognitive function will be evaluated in terms of level of orientation, memory, and concentration (SOMCT). The SOMCT evaluation is performed by requesting the subjects' to recall the current year and month, one sentence, and to repeat in both numerical and reverse order the sequence of the months through the year. These 6 variables yield scores ranging from 0 to 28, with higher scores indicating better cognitive function (Appendix 2).

Subjects will be premedicated with 0.5 to 2 mg midazolam IV in the pre-operative holding area. The subject will be transported to the operating room and assisted onto the operating table, and ASA standard monitoring will be applied as determined by the anesthesiologist and must include an oxygen saturation monitor and bispectral index (BIS) monitor. The BIS monitor will be applied prior to the induction of anesthesia. Subject vital signs and BIS values will be recorded every 5 minutes throughout the operation and recorded on the anesthesia record. The subject will be preoxygenated using spontaneous mask ventilation at 100% fraction of inspired oxygen inspired oxygen fraction (FiO2) and a fresh gas flow of 6 L/min of oxygen for one to four minutes prior to induction. Anesthesia induction will be performed via bolus injection of 2 mg/kg IV propofol and 1 to 2 mcg/kg of fentanyl intravenous (IV) bolus. After completion of bolus injection of propofol, the inhaled anesthetic vaporizer will be opened to 1 MAC (5.4 to 7.4% for desflurane and 1.4 to 2.5% for sevoflurane) based on study randomization for one to two minutes using masked ventilation. Following the masked ventilation a jaw thrust maneuver will be performed, the fresh gas inflow (not vaporizer) will be turned off, and a lubricated LMA will be inserted. The size and brand of of LMA will be recorded. After verification of proper placement and a seal around the LMA, the inflow will be immediately turned back to 4 to 6 L/min of 100% oxygen with the vaporizer set at 1 MAC for three minutes and the patient will be placed on volume or pressure control mechanical ventilation. Ventilation will be verified via documentation of bilateral breath sounds and chest rise. Following three to five minutes, the inhalational anesthesia will be maintained with either desflurane or sevoflurane (0.5 to 1 MAC) inspired in a 50:50 air/oxygen mixture at a total gas flow rate of 1 L/min. This will be based on the randomization of the subject prior to surgery to one of the two groups of inhaled anesthetics. Additional boluses of fentanyl, propofol, or vasopressors will be administered as needed to maintain analgesia and hemodynamics, including heart rate, spontaneous respiratory rate, and mean arterial pressure (MAP), within 20% of baseline. At end of procedure, upon closure of surgical incision, inhalational anesthetic agents will be discontinued and fresh gas flow will be increased to 6 to 8 L/min of 100% oxygen. All patients will be maintained with inhaled anesthestic that will not be below 0.5 MAC for either desflurane or sevoflurane throughout the surgery.

Each episode of coughing during induction of anesthesia until the subject is awake and oriented will be recorded by a blinded observer and graded according to the scale below Coughing is defined as; 1 if a single cough occurred and oxygen saturation (SpO2) ≥ 95 %; 2 if multiple coughs occurred and SpO2 ≥ 95 %; 3 if multiple coughs occurred and SpO2 < 95 %; 4 if multiple coughs occurred, SpO2 < 95 % and coughing requires administration of an IV medication.

Awakening from anesthesia (eye-opening) will be assessed by the research staff by asking the subjects to follow verbal commands only (no touch) at one-minute intervals after the discontinuation of volatile anesthetics. The time to appropriateness for extubation will also be recorded in one-minute intervals after discontinuation of the inhalational agent. Prior to removal of the LMA, the subject will be determined to be awake by "eyes-open" to command and deemed appropriate by the anesthesiologist.

Anesthesia and procedure start and end time, admission and discharge time to the post-anesthesia care unit (PACU) and time to discharge from the hospital will also be recorded.

Post-anesthesia recovery (physical status) will be evaluated, according to the Aldrete score16, 5 minutes after extubation and every 5 minutes until the subject reaches an Aldrete score ≥ 9. Subjects should be able to move the extremities spontaneously or on command, to breathe and cough, have systolic blood pressure values within 20 mmHg of the pre-anesthetic levels or baseline levels, alert or arousable to quiet voice, and able to maintain SpO2 > 90 % with supplementary O2 administration through a face mask at the lowest concentration needed to ensure Pao2 between 100 and 200 mmHg (Appendix 1) After subjects have reached a postoperative Aldrete score ≥9, the research staff will perform a SOMCT test to evaluate postoperative cognitive function every 15 minutes for the first hour after surgery and at the time of discharge from the PACU.

At 24 hours after surgery overall satisfaction will be assessed by asking the subjects about their experience with the anesthetic medication using a 3 point rating scale, by personal interview or phone call, by a blinded research staff. Satisfaction will be rated on a scale: 2 being equivalent to highly satisfied, 1 being equivalent to satisfied and 0 being equivalent to dissatisfied.

All medications taken in the 24 hours prior to treatment will be recorded. Any drug with potential antiemetic properties, intraoperative medication, and daily consumption of opioids will be recorded for 24 hours postoperatively or until discharge from the hospital or whichever comes first. Adverse events and serious adverse events will be recorded from time of consent until discharge.

Safety Assessments:

Safety parameters will be assessed by monitoring vital signs, adverse events, and either urine or serum pregnancy test. A physical exam will be performed at screening.

The occurrence of adverse events (AE) and serious adverse events (SAE) will be recorded from time to consent until discharge. For each adverse event, the relationship to the study medication, severity, expectedness of an adverse event and outcome will be determined by the principal investigator and recorded in the study source accordingly.

In the case a subject withdraws from the study because of a serious adverse event (SAE), the local Institutional Review Board (IRB) will be notified within 10 days.

Adverse event definition

An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject who has been administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign, symptom, abnormal laboratory finding, or a temporal disease associated with the use of a study drug, whether or not considered related to the study drug.

Planned hospital admissions and/or surgical operations for an illness or disease that existed before the subject was enrolled in a clinical study are considered part of the subjects' medical history and are not to be considered AEs.

Serious adverse event

A SAE is any untoward medical occurrence that at any dose:

* Results in death
* Is life-threatening
* Results in persistent or significant disability/incapacity
* Requires in-subject hospitalization or prolongs hospitalization
* Is a congenital anomaly/birth defect
* Is another medically-significant event that, based upon appropriate medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above

Withdrawal criteria from the study

According with the Declaration of Helsinki, participants have the right to withdraw from the study at any time for any reason. The principal investigator also has the right to remove a subject from the study. Reasons for which a subject may be removed from the study include:

* An adverse event
* The request of the subject, his/her legal representative or caregiver, investigator, whether for administrative or any other reasons
* Non - compliance with medication, protocol violation or unreliable, behavior
* Any clinically significant abnormal laboratory values or other clinically significant abnormalities identified by the principal investigator according to his clinical judgment. These will be followed by appropriate tests and/or procedures until these values have returned to normal, to clinically acceptable levels, or can be attributed to other causes other than study drug

The principal investigator may withdraw an enrolled and treated subject from the study for any of the following reasons:

* Occurrence of a serious or intolerable adverse event
* Emergence of a clinically significant change in a laboratory parameter(s)
* The subject requests to be discontinued from the study
* A protocol violation sufficiently serious as to require subject withdrawal
* General or specific changes in the subject's condition that render further treatment unreasonable or unsafe within the standards of clinical practice in the judgment of the principal investigator or treating physician.

Any subject may leave the study at any time. If the subject decides to stop participating in the study, there will be no penalty. The subjects will not lose any benefits to which they are otherwise entitled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 50 to 75 years of age.
2. Subjects with an American Society of Anesthesiologist (ASA) physical status of I to III.
3. Subjects able to provide written informed consent to participate in the study.
4. Female subjects who have a negative urine or serum pregnancy test, who have been surgically sterilized, or are postmenopausal.
5. Subjects scheduled for urological cystoscopic surgery under general anesthesia with LMA intubation.

Exclusion Criteria:

1. Subjects who are prisoners.
2. Subjects who have limited decision-making capacity or lack the ability to consent.
3. Subjects with a history of alcohol or drug abuse within the last year.
4. Subjects with a history of an allergic reaction, intolerance, or contraindications to any of the study medications.
5. Females who are pregnant or are breastfeeding.
6. Subjects with BMI greater than 35.
7. Subjects with a history of hiatal hernia or gastroesophageal reflux disease (GERD).
8. Subjects with a history of pharyngeal pathology.
9. Subjects who have participated in or are currently participating in a clinical trial of an investigational drug within 30 days prior to surgery.
10. Subjects with a fixed decreased pulmonary compliance, such as patients with pulmonary fibrosis.
11. Subjects with multiple or massive injuries, acute abdominal and/or thoracic injuries.
12. Subjects with any condition associated with delayed gastric emptying.
13. Subjects who are profoundly unconscious and who may not resist LMA insertion or have a contraindication for the use of LMA intubation.
14. Subjects with any condition that in the opinion of the investigator would render the subject ineligible for participation in the study, such as unstable or severe cardiovascular, pulmonary, renal, hepatic, metabolic, or endocrine disease or neuromuscular disorder.
15. Subjects with a history of malignant hyperthermia.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Werner, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were approached for consent and were given ample time to decide on participation in the study. This process began in September 2010 and ended in October 2012. All study activity occurred in the hospital or patient clinic.
Pre-assignment Details: Enrolled patients were excluded from group assignments if it was discovered after consent an eligibility criteria was not met. After consent patients were further examined for study eligibility and were excluded if they were unable to recieve LMA for the procedure or had a medical condition which was contraindicated with one of the methods.
Groups:
- Desflurane: Comparing the effect on recovery time in patients undergoing urological cytoscope surgery under general anesthesia with a laryngeal mask airway (LMA) using Desflurane.
  Desflurane : 5.4 to 7.4% desflurane
- Sevoflurane: Comparing the effect on recovery time in patients undergoing urological cytoscope surgery under general anesthesia with a laryngeal mask airway (LMA) using Sevoflurane.
  Sevoflurane : 1.4 to 2.5% Sevoflurane
Period: Overall Study
Arm/Group | Desflurane | Sevoflurane
Started | 38 | 37
Completed | 34 | 32
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Desflurane: Comparing the effect on recovery time in patients undergoing urological cytoscope surgery under general anesthesia with a laryngeal mask airway (LMA) using Desflurane (5.4 to 7.4%)
- Sevoflurane: Comparing the effect on recovery time in patients undergoing urological cytoscope surgery under general anesthesia with a laryngeal mask airway (LMA) using Sevoflurane (1.4 to 2.5%).
- Total: Total of all reporting groups
Arm/Group | Desflurane | Sevoflurane | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (7.7) | 61.3 (6.6) | 61.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 22 | 18 | 40
Region of Enrollment [Number; unit: participants]
  United States | 38 | 37 | 75

OUTCOME MEASURES:

1. Primary Outcome: Recovery Time
Description: Recovery Time after exposure to desflurane or sevoflurane considering time of emergence from anesthesia
Time Frame: 14 Days
Population: Determined if patients passed all eligibility and completed study.
Measure: Median (Inter-Quartile Range); unit: Minutes
Groups:
- Desflurane: Comparing the effect on recovery time in patients undergoing urological cytoscope surgery under general anesthesia with a laryngeal mask airway (LMA) using Desflurane.
  Sevoflurane : 1.4 to 2.5% Sevoflurane
- Sevoflurane: Comparing the effect on recovery time in patients undergoing urological cytoscope surgery under general anesthesia with a laryngeal mask airway (LMA) using Sevoflurane.
  Desflurane : 5.4 to 7.4% desflurane
Arm/Group | Desflurane | Sevoflurane
Number analyzed (Participants) | 34 | 32
Minutes | 9 [5 to 18] | 20 [9 to 27]

2. Secondary Outcome: Difference in Time to Orientation
Description: Difference in time to orientation as measured by Short Orientation Memory Concentration Test (SOMCT) between the desflurane group and the sevoflurane group
Time Frame: 14 Days
Population: Determined if patient passed eligibility and completed study.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Desflurane | Sevoflurane
Number analyzed (Participants) | 34 | 32
Minutes | 15 [5 to 30] | 15 [5 to 30]

3. Secondary Outcome: Time to Extubation
Description: Time from gas discontinuation to eye extubation after eye opening
Time Frame: 14 days
Population: Determined if patient passed eligibility and completed study.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Desflurane | Sevoflurane
Number analyzed (Participants) | 34 | 32
Minutes | 5.0 (2.5) | 7.9 (4.1)

4. Secondary Outcome: Incidence of Coughing at Extubation, Approximately 10 Minutes After End of Surgery
Description: Effect of desflurane versus sevoflurane on the incidence of coughing at extubation using a standardized coughing scale
Time Frame: At extubation, approximately 10 minutes after end of surgery
Population: Determined if patient passed eligibility and completed study.
Measure: Count of Participants; unit: Participants
Arm/Group | Desflurane | Sevoflurane
Number analyzed (Participants) | 34 | 32
Participants | 10 | 4

ADVERSE EVENTS:
Arm/Group | Desflurane | Sevoflurane
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/37
Other Adverse Events (participants affected / at risk) | 12/38 | 4/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desflurane (N=38) | Sevoflurane (N=37)
Coughing (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 4 (4)

LIMITATIONS AND CAVEATS:
Nine patients which were screen failures and not included in final analysis. Patients assessed for SOMCT score every 15 minutes in the PACU, which did not allow for an exact time for the return to cognition endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No